CLINICAL TRIAL: NCT02401711
Title: How Should Surgical Residents Be Educated About Patient Safety in the Operating Room: a Pilot Randomized Trial
Brief Title: How Should Surgical Residents Be Educated About Patient Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, KuoJen Tsao, Associate Professor & The Children's Fund, Inc. Distinguished Professorship in Pediatric Surgery, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HSC-MS-14-0073
Record Dates: First submitted 2015-03-23; First posted 2015-03-30 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Medical Education; Patient Safety; Educational Safety Curriculum; Surgical Resident

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Online training (Active Comparator): Residents randomized to the control group will only participate in the Breakthroughs in Patient Safety (BIPS) online training (Education - BIPS course). All residents in the comparison arm will receive evaluations on their non-technical skills, but the results will not be fed back to them until after the study has been completed.
  Interventions: Behavioral: Education - BIPS course
- Online training & Safety curriculum & Evaluation and feedback (Experimental): Those in the intervention group will participate in a formal safety education curriculum in addition to the currently required Breakthroughs in Patient Safety (BIPS) online training. The intervention will have three components: (1) the mandatory online BIPS course (Education - BIPS course), (2) the formal safety curriculum, and (3) ongoing evaluation and feedback of operating room performance.
  Interventions: Behavioral: Education - BIPS course; Behavioral: Formal safety curriculum; Behavioral: Ongoing evaluation and feedback

INTERVENTIONS:
Behavioral: Education - BIPS course — The guiding principles behind the BIPS program include: (1) explaining how complex systems cause human error and how human error can lead to patient harm in complex systems; (2) diagnosing human error and identifying a prevention behavior for each of the three types: skill, rule, and knowledge; and (3) preventing error by promoting safety behaviors, such as having attention to detail, communicating clearly, having a questioning attitude, and speaking up for safety
Behavioral: Formal safety curriculum — The educational program is designed to improve patient safety by informing residents about safe operating room behaviors.
  Arms: Online training & Safety curriculum & Evaluation and feedback
Behavioral: Ongoing evaluation and feedback — The feedback program is designed to encourage the use of safe behaviors and to discourage unsafe behaviors taught in the workshops.
  Arms: Online training & Safety curriculum & Evaluation and feedback

SUMMARY:
The purpose of this study is to compare the effectiveness of two methods, safety curriculum in addition to online training alone, for teaching patient safety to surgery residents. Despite multiple studies evaluating educational safety curricula, the best methods for teaching residents about patient safety is unknown. It is hypothesized that empowering surgery residents to actively engage in behaviors to increase patient safety may lead to a higher quality perioperative care and communication.

ELIGIBILITY:
Inclusion Criteria:

* All surgery residents at the University of Texas Health Science Center at Houston, from post-graduate year (PGY)-1 to PGY-5.

Exclusion Criteria:

* Non-surgery residents at the University of Texas Health Science Center at Houston.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2014-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Changes in safety culture as measured by the Safety Attitudes Questionnaire (SAQ) | Baseline, One year

SECONDARY OUTCOMES:
Learner satisfaction, knowledge, and behaviors as measured by the Oxford Non-Technical Skills (NOTECHS) system | One year